CLINICAL TRIAL: NCT06114667
Title: Nasal High Flow in Early Management of Patients Admitted to the Emergency Department for Acute Exacerbation of Chronic Obstructive Pulmonary Disease With Hypercapnic Acidosis : a Randomized Controlled Non Inferiority Study
Brief Title: Nasal High Flow Versus Non-invasive Ventilation for Early Treatment of Acute Exacerbation of Chronic Obstructive Pulmonary Disease With Hypercapnic Acidosis
Acronym: HiCOPD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL19_0626; 2022-A02633-40 (Registry Identifier: National Agency for the Safety of Medicines and Health Products)
Record Dates: First submitted 2023-09-04; First posted 2023-11-02 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Acute Exacerbation of Chronic Obstructive Pulmonary Disease; Hypercapnic Acidosis; Respiratory Failure With Hypercapnia
Keywords: respiratory insufficiency; Hypercapnic Acute Respiratory Failure; chronic obstructive pulmonary disease exacerbation; nasal high flow; non invasive ventilation; emergency department; critical are
MeSH Terms: conditions — Acidosis, Respiratory; Respiratory Insufficiency; Emergencies

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either one of two groups of respiratory support (NIV or nasal high flow) in parallel. Randomization will be in a 1:1 ratio, and stratified by center, severity of hypercapnia and acidosis
Masking Description: Masking non feasible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nasal high flow (Experimental): Nasal high flow will be administered through a heated humidifier (Airvo 3, Fisher and Paykel healthcare) and applied through large bore binasal prongs.
  Initial gas flow rate will be set at 60 l/min, FiO2 will be adjusted to maintain an SpO2 88-92% and Initial temperature will be set at 37° and reduced according to patient's tolerance.
  Ventilatory support will be applied in 2h sessions and resumed as needed according to international guidelines for NIV treatment
  Interventions: Device: Ventilatory support via nasal high flow
- Non invasive ventilation (Active Comparator): NIV will be delivered through a face mask connected to a ventilator with pressure support applied in a noninvasive ventilation mode.
  The Pressure-support level will be adjusted to obtain an expired tidal volume of 6-8 ml/kg of predicted body weight and a respiratory rate of 25-30 b/min. PEEP (range 5-10 cm of water) and FiO2 will be adjusted to maintain an SpO2 88-92% and to patient's comfort.
  Ventilatory support will be applied in 2h sessions and resumed as needed according to international guidelines for NIV treatment.
  Interventions: Device: Ventilatory support via NIV

INTERVENTIONS:
Device: Ventilatory support via nasal high flow — Ventilatory support will be applied in 2h sessions and resumed as needed according to international guidelines for NIV treatment.
  Arms: Nasal high flow
Device: Ventilatory support via NIV — Ventilatory support will be applied in 2h sessions and resumed as needed according to international guidelines for NIV treatment.
  Arms: Non invasive ventilation

SUMMARY:
The purpose of this study is to determine whether nasal high flow is non inferior to non invasive ventilation (NIV) in the early treatment of patients with acute exacerbation of chronic obstructive pulmonary disease (AE-COPD) and hypercapnic acidosis in the emergency department (ED). After obtaining informed consent, participants will be randomly assigned to receive either nasal high flow or non invasive ventilation (NIV, reference treatment) as respiratory support. Researchers will compare both respiratory support groups to see if their blood gas analysis and respiration return to normal ranges.

DETAILED DESCRIPTION:
Prospective multicenter comparative therapeutic study, with a randomized controlled parallel and open design. Nasal high flow will be compared to NIV (reference treatment) for early treatment of AE-COPD associated with hypercapnic acidosis.

Adult patients admitted to the ED for AE-COPD with hypercapnic acidosis will be randomized to receive either nasal high flow or NIV as ventilatory support. Ventilatory support will be applied in 2h sessions and resumed as needed according to international guidelines for NIV treatment. Close monitoring of clinical and gas parameters will be conducted with repeat assessment and serial blood gas testing at 2h and after each 2h session of respiratory support in the ED (2h, 4h, 6h) and at 24h.

Standard oxygen therapy will be administered as required between ventilatory support sessions to maintain a target peripheral oxygen saturation (SpO2 : 88-92%).

Patient's dyspnea and comfort will be assessed before treatment and at 2h, and after each respiratory support session in the ED Patients will receive standard medical treatment for AE-COPD (bronchodilator, corticosteroids and antibiotics) according to current practice and 2023 global initiative guidelines for the management of COPD (GOLD).

Patients will be followed up at day 28 by means of medical records review and telephone interview

ELIGIBILITY:
Adult Patient admitted to the ED for acute exacerbation of COPD (AE-COPD)and respiratory acidosis (PaCO2 > 45 mmHg and pH <7.35), for whom ventilatory assistance by NIV is indicated (SPLF 2017, GOLD2023 recommendations)

Inclusion Criteria:

* Patients with ability to understand and give an informed consent
* Patients affiliated with or who benefit from a social security
* Patients admitted to the emergency department for a clinical suspicion of AE-COPD based on clinical history, physical examination and chest X-ray (SPLF 2017)
* Patients with acute respiratory failure defined by: Respiratory rate ≥ 25 bpm AND/OR Signs of respiratory failure (use of accessory respiratory muscles, paradoxical abdominal movement)
* Patients with respiratory acidosis defined by PaCO2 > 45 mmHg AND pH < 7.35 (measured on arterial blood gas)

Exclusion Criteria:

* Patients who have already received NIV treatment before inclusion (including in-hospital or prehospital, with the exception of NIV at home)
* Contraindication to non-invasive ventilation (SPLF 2017 and GOLD 2023 recommendations)
* Patient uncooperative, agitated, opponent of the technique

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in PaCO2 | 2 hours
  PaCO2 will be measured from standard laboratory arterial blood gas analysis before the initiation of ventilatory assistance and after 2 hours of treatment

SECONDARY OUTCOMES:
Change in pH | 2 hours
  Blood gas parameters will be measured from standard laboratory arterial blood gas analysis before the initiation of ventilatory support and after 2 hours of treatment
Change in PaO2 | 2 hours
  Blood gas parameters will be measured from standard laboratory arterial blood gas analysis before the initiation of ventilatory support and after 2 hours of treatment
Change in PaCO2 | up to 24 hours
  Blood gas parameters will be measured from standard laboratory arterial blood gas analysis before the initiation of ventilatory support and after sessions of ventilatory support
Change in pH | up to 24 hours
  Blood gas parameters will be measured from standard laboratory arterial blood gas analysis before the initiation of ventilatory support and after sessions of ventilatory support
Change in PaO2 | up to 24 hours
  Blood gas parameters will be measured from standard laboratory arterial blood gas analysis before the initiation of ventilatory support and after sessions of ventilatory support
Respiratory rate | up to 24 hours
  Clinical parameters will be monitored by physician at baseline and throughout ventilatory support sessions, according to the international guidelines for NIV monitoring
Signs of increased work of breathing (use of accessory respiratory muscles, paradoxical motion of the abdomen) | up to 24 hours
  Use of accessory respiratory muscles and paradoxical motion of the abdomen will be assessed by physician at baseline and after sessions of ventilatory support, on a 5 point likert scale (from 1 : absence to 5 : maximal use or accessory respiratory muscle and paradoxical motion of the abdomen)
Perceived dyspnea | up to 24 hours
  Dyspnea will be assessed by the patient using a Modified Borg scale for dyspnea, at baseline and after sessions of ventilatory support. Difficulty of breathing will be quantified on a scale from 0 : no difficulty at all to 10 : breathing difficulty is maximal.
Treatment failure (composite of change of treatment arm / need for invasive mechanical ventilation/ mortality) | Up to Day 28
  Failure will be defined by a composite of clinical or gasometric worsening or patient intolerance inducing a change of treatment arm/ need for orotracheal intubation and/or mortality (all causes).
Weaning from ventilatory support | Up to Day 28
  Delay from initiation of ventilatory support to weaning

OTHER OUTCOMES:
Hospitalization rate, including hospitalization in critical care units | Day 28
  Proportion of patients requiring hospitalization following ED management
Readmission for AE-COPD | Day 28
  Proportion of patients requiring emergency department admission for AE-COPD within 28 days from index admission

CONTACTS AND LOCATIONS:
Overall Officials: Mustapha Sebbane, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (3):
- France (3):
  - Centre hospitalier universitaire de Montpellier, Montpellier
  - Centre hospitalier universitaire de Nimes, Nîmes
  - Centre Hospitalier Universitaire de Poitiers, Poitiers

IPD SHARING:
Plan to Share IPD: Undecided